CLINICAL TRIAL: NCT01725945
Title: A Pilot Study of the DASH Diet in Not-Well-Controlled Adult Asthma
Brief Title: The DASH Diet for Adults With Uncontrolled Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Medical Foundation (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Kaiser Permanente (Other); Stanford University (Other)
Responsible Party: Principal Investigator, Jun Ma, MD, PhD, Associate Investigator, Palo Alto Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R34HL108753 (NIH); R34HL108753 (NIH)
Record Dates: First submitted 2012-11-07; First posted 2012-11-14 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Asthma; Hypertension
Keywords: DASH; diet; asthma; adults; asthma control
MeSH Terms: conditions — Asthma; Hypertension

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): Usual Care
- DASH Intervention (Experimental): Dietary Approaches to Stop Hypertension dietary pattern. Usual care in combination with a DASH intervention consisting of 8 group and 3 individual sessions over 3 months, followed by 3 monthly phone consultations.
  Interventions: Behavioral: Dietary Approaches to Stop Hypertension dietary pattern

INTERVENTIONS:
Behavioral: Dietary Approaches to Stop Hypertension dietary pattern — The intervention will employ a series of small group and individual sessions, followed by periodic telephone contacts, to help participants make appropriate dietary changes and develop the skills to maintain these changes over the long term. The initial 3 months of intensive intervention will involve 8 group and 3 individual sessions for 45-60 minutes each. During the next 3 months, participants will receive counseling phone calls once per month for 20-30 minutes each call. Group session sizes may range from 8-15 participants.
  Other Names: DASH
  Arms: DASH Intervention

SUMMARY:
Dietary intervention efficacy trials are distinctly lacking in asthma research. This pilot study aims to provide effect size estimates and justification, clinical trial and intervention feasibility data, and procedural materials for a full-scale randomized controlled trial that will determine the efficacy and mechanisms of action of the Dietary Approaches to Stop Hypertension (DASH)-a recommended dietary pattern based on proven cardiovascular benefits-as adjunct therapy to standard care for adults with uncontrolled asthma.

DETAILED DESCRIPTION:
Dietary intervention efficacy trials are distinctly lacking in asthma research. This pilot study aims to provide effect size estimates and justification, clinical trial and intervention feasibility data, and procedural materials for a full-scale randomized controlled trial that will determine the efficacy and mechanisms of action of the Dietary Approaches to Stop Hypertension (DASH)-a recommended dietary pattern based on proven cardiovascular benefits-as adjunct therapy to standard care for adults with uncontrolled asthma. Eligible, consenting participants (n=90) will be randomized to receive usual care alone or combined with a DASH intervention. Follow-up assessments will occur at 3 and 6 months. By evaluating a dietary pattern approach to improving asthma control, this study could advance the evidence base for refining clinical guidelines and public health recommendations regarding the role of dietary modifications in asthma management.

ELIGIBILITY:
Inclusion Criteria:

* Ethnicity: All ethnic groups
* Body mass index (BMI) 18.5-39.9 kg/m2
* Suboptimally controlled asthma:
* Diagnosis of asthma on the current medical problem list
* Currently prescribed at least 1 medication for the treatment of asthma
* Physiological evidence of asthma with demonstrable reversibility of airway obstruction, or a specialist's confirmation of asthma diagnosis based on chart review
* Documented history of high asthma-related emergency and/or inpatient encounters or reliever medication usage
* Asthma Control Test: total score <20 or item score <3 for any of the first 4 questions regarding symptoms (3-6x/week or more), nighttime awakening (1x/week or more), interference with normal activity (at least some of the time), and rescue medication use for symptom relief (2-3x/week or more)
* Kaiser member for ≥1 year
* PCP approval of study screening
* Able and willing to enroll and provide written informed consent

Exclusion Criteria:

* Intermittent asthma, defined as either seasonal asthma or (daytime asthma symptoms <2x/week and nocturnal symptoms <2x/month and no use of long-term control medications)
* Primary diagnosis of COPD (emphysema or chronic bronchitis) on the current medical problem list or suggested by baseline spirometry and smoking history
* Previous diabetes (other than during pregnancy) or diabetes diagnosed as a result of fasting blood glucose or hemoglobin A1c levels obtained at screening
* Previous cardiovascular disease: e.g., coronary heart disease, cerebrovascular disease, peripheral vascular disease, heart failure, or aortic aneurysm
* Diagnosis of cancer (other than non-melanoma skin cancer) that is/was active or treated with radiation or chemotherapy within the past 2 years
* Inflammatory bowel disease, colostomy, malabsorption, or major gastrointestinal resection
* Diagnosis of bipolar or psychotic disorder or hospitalization for psychological or emotional problems within the last 2 years
* Diagnosis of a terminal illness and/or in hospice care
* Fasting LDL cholesterol >190 mg/dL, triglycerides >500 mg/dl, fasting blood glucose >125 mg/dl
* Significant liver enzyme abnormality as indicated by AST or ALT more than 2 times the upper limit of normal or a clinical diagnosis of hepatitis
* Renal insufficiency (GFR<60 ml/min)
* Current use of insulin or oral hypoglycemic agents
* Use of oral corticosteroids >5 days/month on average
* Current use of medications for treatment of psychosis or manic-depressive illness
* Current use of prescription or non-prescription weight-loss products or any dietary/herbal supplements and unwillingness to discontinue;
* Inability to speak, read, or understand English at the 6th-grade level or above
* Inability to perform pulmonary function tests by spirometry in a consistent manner
* DASH concordance index >60%
* Unwillingness to modify current diet
* Current or planned participation in a structured program that overtly focuses on diet and nutrition
* Planning to undergo bariatric surgery during the study period
* Actively attempting to lose weight, or weight change >15 lbs during prior 3 months
* Consumption of >21 alcoholic drinks per week, or >=6 drinks on one occasion twice or more per week, or alcoholism as determined by the Alcohol Use Disorders Identification Test
* Pregnant, lactating, or planning to become pregnant during the study period
* No longer a Kaiser patient or planning to transfer care out of Kaiser or to move out of the area during the study period
* Family/household member of another study participant or of a study staff member
* Enrolled or planning to enroll in another research study that would limit full participation in the study or confound the interpretation of the study's findings
* Investigator discretion for safety or protocol adherence reasons

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
7-item Juniper Asthma Control Questionnaire (ACQ) | 6-months post-randomizaton
  The ACQ provides a reliable, validated assessment of asthma control focusing on current impairment. Its 7 items assess the components of current asthma impairment as defined in the asthma treatment guidelines, i.e., daytime and nocturnal asthma symptoms, activity limitations, rescue medication use (excluding use to prevent exercise-induced bronchospasm), and lung function (FEV1). The ACQ is the only guideline-recommended composite measure of asthma control that includes lung function in its overall rating.

SECONDARY OUTCOMES:
Lung function | 6-months post-randomization
  Lung function measured by spirometry
Asthma specific Quality of Life | 6-months post-randomization
  Juniper Mini Asthma Quality of Life Questionnaire (Mini-AQLQ)
Asthma symptom-free and β2-agonist-free days | 6-months post-randomization
  Asthma symptom-free and β2-agonist-free days will be calculated from 2-week asthma symptom diaries.
Asthma-related health care utilization | 6 months pre-and post-randomization
  Asthma-related health care utilization will be assessed through data extraction from Kaiser Permanente (KP) electronic databases for the periods of 6 months pre- and post-randomization
Diet adherence | 6-months post-randomization
  Participants' adherence to the DASH diet will be assessed by multiple-pass 24-hour diet recalls for servings of fruits, vegetables, dairy products, and whole grains; increases in serum carotenoids, folate and vitamin B12; and reductions in fasting plasma lipids.
Psychosocial predictors of dietary change | 6-months post-randomization
  Self-efficacy and social support for dietary change will be assessed using previously validated instruments.
Comorbidities | 6-months post-randomization
  Sleep apnea and gastroesophageal reflux disease (GERD) are common comorbidities of obesity and asthma. The Berlin Questionnaire for Sleep Apnea and the GERD Symptom Assessment Scale will be administered to screen for these conditions and to assess changes in symptoms. In addition, the Pittsburgh Sleep Quality Index will be used to assess participants' usual sleep habits and sleep quality. The 9-item Patient Health Questionnaire (PHQ-9) is both a measure of depressive symptomatology and a tentative diagnostic instrument for the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) depressive disorders.
Generic health related Quality of Life | 6-months post-randomization
  The 12-item Short Form Health Survey (SF-12) is a widely used measure to assess non-disease specific physical and mental health status.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, MD, PhD, Principal Investigator — Palo Alto Medical Foundation
Locations (2):
- United States (2):
  - Kaiser Permanente, Hayward Medical Center, Allergy Department, Hayward, California
  - Kaiser Permanente, San Francisco Medical Center, Allergy Department, San Francisco, California

REFERENCES:
- [Derived] Nygaard UC, Xiao L, Nadeau KC, Hew KM, Lv N, Camargo CA, Strub P, Ma J. Improved diet quality is associated with decreased concentrations of inflammatory markers in adults with uncontrolled asthma. Am J Clin Nutr. 2021 Sep 1;114(3):1012-1027. doi: 10.1093/ajcn/nqab063. PMID 33871602
- [Derived] Lv N, Xiao L, Camargo CA Jr, Wilson SR, Buist AS, Strub P, Nadeau KC, Ma J. Abdominal and general adiposity and level of asthma control in adults with uncontrolled asthma. Ann Am Thorac Soc. 2014 Oct;11(8):1218-24. doi: 10.1513/AnnalsATS.201405-214OC. PMID 25343191
- [Derived] Ma J, Strub P, Lavori PW, Buist AS, Camargo CA Jr, Nadeau KC, Wilson SR, Xiao L. DASH for asthma: a pilot study of the DASH diet in not-well-controlled adult asthma. Contemp Clin Trials. 2013 Jul;35(2):55-67. doi: 10.1016/j.cct.2013.04.008. Epub 2013 May 3. PMID 23648395